CLINICAL TRIAL: NCT01371045
Title: Hormonal and Metabolic Responses to Oral Glucose During Somatostatin Analog Use
Brief Title: Oral Glucose Tolerance Testing (OGTT) on Patients Taking Somatostatin Analogs
Status: Withdrawn | Type: Observational
Why Stopped: PI moved from the institution. Study did not enroll any patients.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Odelia Cooper, Professor of Medicine, Cedars-Sinai Medical Center
Other Study IDs: Pro00024880
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Acromegaly
Keywords: Acromegaly; Growth Hormone; Carcinoid Syndrome; Somatostatin
MeSH Terms: conditions — Acromegaly; Serotonin Syndrome | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood will be drawn (approx. 64cc) to gather baseline hormone and metabolic panels. Blood will again be collected (approx. 36cc) during the Oral Glucose Tolerance Test.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acromegaly: Patients carrying the diagnosis of acromegaly who are on long-acting somatostatin for at least 3 months prior to study enrollment.
  Interventions: Other: Oral Glucose Tolerance Test (OGTT)
- Carcinoid Syndrome: Patients carrying a diagnosis of carcinoid syndrome who are taking long-acting somatostatin for at least 3 months prior to study enrollment.
  Interventions: Other: Oral Glucose Tolerance Test (OGTT)
- Healthy Controls
  Interventions: Other: Oral Glucose Tolerance Test (OGTT)

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — An OGTT is a test that lowers growth hormone in the body to very low levels for a short time in order to see how low the growth hormone levels are in your blood.

SUMMARY:
The purpose of this study is to test the effect of long-acting somatostatin analog medications, taken by patients with acromegaly or carcinoid syndrome, on growth hormone in comparison to healthy controls who are not receiving the medication in order to see whether or not the medication makes the oral glucose test less accurate. The Oral Glucose Tolerance Test (OGTT) is a standard test to measure growth hormone secretion. By comparing GH responses in non-acromegaly subjects taking somatostatin analog treatment, the relative contribution of the medication and the underlying disease state can be analyzed.

DETAILED DESCRIPTION:
Subjects will be informed of the study and after providing written informed consent, subjects will be asked to undergo a 2-hour oral glucose tolerance test (ingestion of 75g glucose with subsequent timed assessment of growth hormone, glucose, insulin and related binding proteins.) Baseline assessment of hormones that may contribute to the results will be drawn, prior to performing the test. Patients will be asked to complete one visit total to participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly or carcinoid syndrome
* Treatment with somatostatin analog therapy (must have established a stable dose of three or more injections on the same dose prior to study enrollment)
* Healthy control subjects

Exclusion Criteria:

* Diagnosis of Diabetes Mellitus (Type 1 or Type 2)
* Use of medication for the treatment of insulin resistance or diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollment will include subjects diagnosed with acromegaly or carcinoid syndrome who are taking long-acting somatostatin analogs for at least three months prior to study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Growth hormone response to OGTT | 2 hours
  assessment of the validity of GH suppression during somatostatin analog treatment in acromegaly and non-acromegaly subjects

CONTACTS AND LOCATIONS:
Overall Officials: Odelia Cooper, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Pituitary Center, Los Angeles, California, United States

REFERENCES:
- [Background] Earll JM, Sparks LL, Forsham PH. Glucose suppression of serum growth hormone in the diagnosis of acromegaly. JAMA. 1967 Aug 21;201(8):628-30. No abstract available. PMID 5006772
- [Background] Giustina A, Chanson P, Bronstein MD, Klibanski A, Lamberts S, Casanueva FF, Trainer P, Ghigo E, Ho K, Melmed S; Acromegaly Consensus Group. A consensus on criteria for cure of acromegaly. J Clin Endocrinol Metab. 2010 Jul;95(7):3141-8. doi: 10.1210/jc.2009-2670. Epub 2010 Apr 21. PMID 20410227
- [Background] Vierhapper H, Heinze G, Gessl A, Exner M, Bieglmayr C. Use of the oral glucose tolerance test to define remission in acromegaly. Metabolism. 2003 Feb;52(2):181-5. doi: 10.1053/meta.2003.50036. PMID 12601629
- [Background] Carmichael JD, Bonert VS, Mirocha JM, Melmed S. The utility of oral glucose tolerance testing for diagnosis and assessment of treatment outcomes in 166 patients with acromegaly. J Clin Endocrinol Metab. 2009 Feb;94(2):523-7. doi: 10.1210/jc.2008-1371. Epub 2008 Nov 25. PMID 19033371
- [Background] Rubeck KZ, Madsen M, Andreasen CM, Fisker S, Frystyk J, Jorgensen JO. Conventional and novel biomarkers of treatment outcome in patients with acromegaly: discordant results after somatostatin analog treatment compared with surgery. Eur J Endocrinol. 2010 Nov;163(5):717-26. doi: 10.1530/EJE-10-0640. Epub 2010 Sep 2. PMID 20813787
- [Background] ROTH J, GLICK SM, YALOW RS, BERSON SA. Secretion of human growth hormone: physiologic and experimental modification. Metabolism. 1963 Jul;12:577-9. No abstract available. PMID 13975314
- [Background] Arafat AM, Mohlig M, Weickert MO, Perschel FH, Purschwitz J, Spranger J, Strasburger CJ, Schofl C, Pfeiffer AF. Growth hormone response during oral glucose tolerance test: the impact of assay method on the estimation of reference values in patients with acromegaly and in healthy controls, and the role of gender, age, and body mass index. J Clin Endocrinol Metab. 2008 Apr;93(4):1254-62. doi: 10.1210/jc.2007-2084. Epub 2008 Jan 2. PMID 18171702